CLINICAL TRIAL: NCT06346756
Title: Clinical Evaluation of Class II Restorations Performed With High-fill Injectable Composite and Condensable Universal Composites
Brief Title: Clinical Evaluation of Class II Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Merve Gurses, Assistant Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SelcukA
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Dental Caries; Dental Caries Class II
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- G-aenial A'CHORD universal composite (Experimental)
  Interventions: Other: Treatment of dental caries.
- Tetric Prime universal composite (Experimental)
  Interventions: Other: Treatment of dental caries.
- Filtek Ultimate universal composite (Experimental)
  Interventions: Other: Treatment of dental caries.
- G-aenial Universal Injectable composite (Experimental)
  Interventions: Other: Treatment of dental caries.

INTERVENTIONS:
Other: Treatment of dental caries. — The researchers used G-aenial Universal Injectable (GCI), G-aenial A'CHORD (GCA), Tetric Prime (TP), and Filtek Ultimate (FU) composites for premolar Class II restorations.

SUMMARY:
This study aims to evaluate the one-year clinical performance of Class II restorations made with high-filling injectable and condensable universal composite resins.

The study included 71 patients and 140 restorations. It used G-aenial Universal Injectable (GCI), G-aenial A'CHORD (GCA), Tetric Prime (TP), Filtek Ultimate (FU) composites, and the Clearfil SE Bond adhesive system. Restorations were evaluated and scored according to modified USPHS criteria at seven days, six months, and one year. Chi-square and Cochran Q tests were used for statistical analysis (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

A patient presenting with;

1. over 18 years of age
2. a normal periodontal status and good general health
3. proximal caries that are similar in size to premolar and molar teeth
4. vital teeth
5. teeth in contact with the opposing tooth and subjected to normal occlusal forces
6. attend follow-up appointments

Exclusion Criteria:

1. poor oral hygiene status
2. those with severe or chronic periodontitis
3. absence of adjacent and antagonist teeth
4. potential behavioral problems (e.g. bruxism)
5. allergy to any product used in the study
6. exposure of the pulp during cavity preparation
7. systemically unhealthy
8. pregnant and lactating women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Retention | seventh day, sixth month, twelfth month
  No loss of restorative material

SECONDARY OUTCOMES:
color match | seventh day, sixth month, twelfth month
  The restoration matches the adjacent tooth structure in color and translucency
marginal adaptation | seventh day, sixth month, twelfth month
  There is no visible evidence of a crevice along the margin into which the explorer will penetrate
marginal discoloration | seventh day, sixth month, twelfth month
  There is no discoloration anywhere on the margin between the restoration and the tooth structure
surface texture | seventh day, sixth month, twelfth month
  The surface of the restoration does not have any defects
anatomical form | seventh day, sixth month, twelfth month
  The restoration is continuous with the existing anatomic form
secondary caries | seventh day, sixth month, twelfth month
  No evidence of secondary caries
postoperative sensitivity | seventh day, sixth month, twelfth month
  No postoperative sensitivity, after the restorative procedure and during the study

CONTACTS AND LOCATIONS:
Overall Officials: Merve Gürses, Principal Investigator — Selcuk University, Faculty of Dentistry
Locations (1):
- Selcuk University, Faculty of Dentistry, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No